CLINICAL TRIAL: NCT00935272
Title: A Randomized, Evaluator-Blinded, No-Treatment-Controlled Study of the Effectiveness and Safety of Restylane® in the Augmentation of Soft Tissue Fullness of the Lips
Brief Title: Safety/Efficacy Study of Restylane® in Lip Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medicis Global Service Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MA-1300-15
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Results first posted 2012-01-30 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2011-12

CONDITIONS: Lip Augmentation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Restylane® Treatment
  Interventions: Device: Restylane®
- Non-Treatment (No Intervention): Non-Treatment Arm
  Interventions: Device: Non-Treatment

INTERVENTIONS:
Device: Restylane® — Restylane® injections in the lips
  Arms: Treatment
Device: Non-Treatment — Non- Treatment
  Arms: Non-Treatment

SUMMARY:
To determine the safety and effectiveness of Restylane® when used for lip augmentation.

ELIGIBILITY:
Inclusion Criteria:

* Must meet established lip fullness criteria

Exclusion Criteria:

* Allergic to injectable hyaluronic acid, local topical anesthetics or nerve blocking agents; Conditions/procedures that could interfere with lip fullness evaluations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Corey, MBA, Study Chair — Medicis Global Service Corporation
Locations (12):
- United States (12):
  - Call for Information, San Diego, California
  - Call for Information, San Francisco, California
  - Call for Information, Santa Monica, California
  - Call for Information, New Haven, Connecticut
  - Call for Information, Coral Gables, Florida
  - Call for Information, Miami Beach, Florida
  - Call for Information, Hunt Valley, Maryland
  - Call for Information, Chestnut Hill, Massachusetts
  - Clinton Twp., Michigan
  - Call for Information, Warren, Michigan
  - Call for Information, Mount Kisco, New York
  - Call for Information, Chapel Hill, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first enrollment: July 20, 2009 Date last subject completed: June 1, 2010 180 subjects enrolled from 12 investigational centers
Pre-assignment Details: Subjects with Fitzpatrick Skin Types I, II or III (lighter skin types) needed both lips to be assessed as very thin or thin to meet enrollment criteria.
  Subjects with Fitzpatrick Skin Types IV, V or VI (darker skin types) need at least one lip to be assessed as very thin or thin to meet enrollment criteria.
Groups:
- Treatment With Restylane: Restylane is composed of a clear, colorless and transparent gel in sterile 1.0 mL syringes. It is supplied with a sterilized 30G x ½ inch needle. The number of syringes used depends on the amount needed to achieve optimal lip augmentation. Optimal lip augmentation is defined as the best possible aesthetic result that can be obtained. Treatment will occur on day 1, with an optional 2 week touch-up at the investigator's and patient's discretion.
- No Treatment: Subjects who received no treatment, for comparison purposes, for the primary efficacy and safety analysis
Period: Overall Study
Arm/Group | Treatment With Restylane | No Treatment
Started | 135 | 45
Completed | 116 | 39
Not Completed | 19 | 6
Not completed — Lost to Follow-up | 10 | 3
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment With Restylane | No Treatment | Total
Number analyzed (Participants) | 135 | 45 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 133 | 44 | 177
  >=65 years | 1 | 1 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 47.8 (10.5) | 47.2 (10.9) | 47.6 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 45 | 179
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 135 | 45 | 180

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response
Description: Assessment of lip fullness augmentation after treatment with Restylane, as compared to no treatment, at week 8 as compared to baseline assessment. Response was determined by at least one grade improvement from baseline in the upper and lower lips using the Medicis Lip Fullness Scale (MLFS). The MLFS is a 5 number scale with grading: (1) Very Thin, (2) Thin (3) Medium (4) Full and (5)Very Full.
Time Frame: Baseline and at 8 weeks
Population: Analysis was ITT; Sample size based upon a one-sided Fisher's Exact test with alpha = 0.05; Subjects with a missing Blinded Evaluator assessment as Week 8 were imputed using the hot deck method
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment With Restylane | No Treatment
Number analyzed (Participants) | 135 | 45
Percentage of Participants | 92.6 [86.8 to 96.4] | 28.9 [16.4 to 44.3]

2. Secondary Outcome: Percentage of Participants With a Response
Description: Assessment of lip fullness augmentation after treatment with Restylane, as compared to no treatment, at post-baseline time points as compared to baseline assessment. Response was determined by at least one grade improvement from baseline in the upper and lower lips using the Medicis Lip Fullness Scale (MLFS). The MLFS is a 5 number scale with grading: (1) Very Thin, (2) Thin (3) Medium (4) Full and (5)Very Full.
Time Frame: Baseline and at weeks 12, 16, 20 and 24
Population: For this secondary objective, the pool of participants analyzed was based on 135 from the Intent to Treat population. However the analysis was done with the number of subjects with non-missing data. This number varied for each timepoint.
Measure: Number (95% Confidence Interval); unit: Percent of responders
Arm/Group | Treatment With Restylane | No Treatment
Number analyzed (Participants) | 135 | 45
Percent of responders
  Week 12 | 90.1 [83.3 to 94.8] | 36.8 [21.8 to 54.0]
  Week 16 | 84.2 [76.4 to 90.2] | 35.9 [21.2 to 52.8]
  Week 20 | 75.0 [66.1 to 82.6] | 33.3 [19.1 to 50.2]
  Week 24 | 69.6 [60.3 to 77.8] | 36.8 [21.8 to 54.0]

ADVERSE EVENTS:
Groups:
- Treatment With Restylane; No Treatment: Safety included post treatment assessment, and assessments at each visit throughout the study.
- Second Treatment: At Week 24, subjects who were initially randomized to treatment were offered an optional second treatment with Restylane. In addition those randomized to non-treatment were offered their first treatment of Restylane at week 24. The safety from this set was followed to one month after the treatment.
Arm/Group | Treatment With Restylane | No Treatment | Second Treatment
Serious Adverse Events (participants affected / at risk) | 4/135 | 1/45 | 0/93
Other Adverse Events (participants affected / at risk) | 149/172 | 5/45 | 60/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With Restylane (N=135) | No Treatment (N=45) | Second Treatment (N=93)
Acute Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Not related to Restylane as determined by the physician.
Transient Ischemic Attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Probably not related to Restylane as determined by the physician.
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Not related to Restylane as determined by the physician.
Streptococcus Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Not related to Restylane as determined by the physician.
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) — Not related to Restylane as determined by the physician.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With Restylane (N=172) | No Treatment (N=45) | Second Treatment (N=93)
Pain (General disorders) | 36 (97) | 1 (1) | 19 (51)
Swelling (General disorders) | 100 (224) | 0 (0) | 52 (103)
Tenderness (General disorders) | 38 (69) | 0 (0) | 16 (29)
Nasopharyngitis (Infections and infestations) | 9 (9) | 2 (3) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 76 (131) | 0 (0) | 26 (41)
Headache (Nervous system disorders) | 12 (17) | 2 (3) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 29 (57) | 0 (0) | 10 (19)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 14 (21) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days